CLINICAL TRIAL: NCT02814409
Title: Alteplase-Tenecteplase Trial Evaluation for Stroke Thrombolysis (ATTEST 2)
Brief Title: Alteplase-Tenecteplase Trial Evaluation for Stroke Thrombolysis
Acronym: ATTEST2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other); University of Edinburgh (Other); Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GN14NE598
Record Dates: First submitted 2016-06-23; First posted 2016-06-27 (Estimated); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Tissue Plasminogen Activator; Tenecteplase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alteplase - standard care (Active Comparator): Alteplase 0.9 mg/kg with 10% of the total dose administered as an initial intravenous bolus and remaining 90% of the total dose administered as an intravenous infusion over 1 hour (maximum dose 90mg).
  Interventions: Drug: Intravenous recombinant tissue plasminogen activator (rtPA) Alteplase
- Tenecteplase (Experimental): Tenecteplase 0.25mg/kg administered as a single rapid intravenous bolus (maximum dose 25mg).
  Interventions: Drug: Intravenous Tenecteplase

INTERVENTIONS:
Drug: Intravenous recombinant tissue plasminogen activator (rtPA) Alteplase — IV Alteplase 0.9mg/kg (max 90mg) bolus + 1h infusion
  Other Names: Actilyse; recombinant tissue plasminogen activator (rtPA)
  Arms: Alteplase - standard care
Drug: Intravenous Tenecteplase — IV Tenecteplase 0.25mg/kg (max 25mg) single bolus
  Other Names: Metalyse; TNK
  Arms: Tenecteplase

SUMMARY:
The principle research question is: in patients with acute ischaemic stroke eligible for intravenous (IV) thrombolysis, is tenecteplase superior in efficacy to alteplase, based on functional outcome as assessed by modified Rankin Scale distribution at day 90?

ELIGIBILITY:
Inclusion criteria:

* Eligible for intravenous thrombolysis.
* Male or non-pregnant female ≥18 years of age.
* <4.5h after symptom onset.
* Consent of patient or legal representative.
* Independent prior to the stroke (estimated modified Rankin Scale 0-2).

Exclusion criteria:

* Eligible for intravenous thrombolysis: Evidence of intracranial haemorrhage or significant non-stroke intracranial pathology likely to account for clinical presentation or represent a risk of intracerebral haemorrhage (eg Central Nervous System neoplasm) on pre-treatment computerised tomography (CT) scan; Stroke within the previous 14 days, thrombolytic therapy within the past 14 days, or hypodensity on pre-treatment computerised tomography (CT) scan consistent with recent cerebral ischaemia other than the presenting event; Systolic blood pressure more than 185 or diastolic blood pressure more than 110 mmHg, or aggressive management (intravenous pharmacotherapy) necessary to reduce blood pressure to these limits; Clinical history suggestive of subarachnoid haemorrhage even if no blood is evident on computerised tomography (CT) scan; High risk of haemorrhage, including major surgery, trauma or gastrointestinal or urinary tract haemorrhage within the previous 21 days; Arterial puncture at a non-compressible site within the previous 7 days; Prolonged cardiopulmonary resuscitation (> 2 minutes) within the previous 14 days; Acute pericarditis and/or subacute bacterial endocarditis; acute pancreatitis; Severe hepatic dysfunction, including hepatic failure, cirrhosis, portal hypertension (oesophageal varices) and active hepatitis; Active peptic ulceration; Known history of haemorrhagic stroke; Known defect of clotting or platelet function (other than antiplatelet therapy); Hypo- or hyperglycaemia (blood glucose <2 mmol/l or >18 mmol/l) sufficient to account for neurological symptoms; Seizure at onset of symptoms unless brain imaging identifies positive evidence of significant brain ischaemia (eg early ischaemic change or hyperdense vessel on plain computerised tomography (CT) scan, computerised tomography angiography (CTA) scan confirmed arterial occlusion); Pregnancy (for women of child-bearing potential a negative pregnancy test will be required prior to randomisation); Inadequate haemostasis: Taking warfarin and international normalised ratio (INR) >1.3, Taking a Direct Oral Anticoagulant (dabigatran, rivaroxaban, apixaban, edoxaban) unless known to be >12 hours since last dose and with normal coagulation assays, Low molecular weight heparin (at doses other than prophylaxis of venous thromboembolism) administered within the preceding 48 hours, Unfractionated heparin administered within the previous 48 hours and activated partial thromboplastin time (APTT) is prolonged.
* Any major medical condition likely to limit survival to day 90.
* Unavailable for day 90 follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1858 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
modified Rankin Scale | Day 90 (+/- 7)
  modified Rankin Scale (mRS) at day 90, determined by the Rankin Focused Assessment (RFA) method using centralised telephone interview, analysed by ordinal distribution ("shift") analysis of the scores in intervention and control groups.

SECONDARY OUTCOMES:
Full neurological recovery (modified Rankin Scale 0-1 versus 2-6). | Day 90 (+/- 7)
  Full neurological recovery (modified Rankin Scale 0-1 versus 2-6).
Independent recovery (modified Rankin Scale score 0-2 versus 3-6). | Day 90 (+/- 7)
  Independent recovery (modified Rankin Scale score 0-2 versus 3-6).
Early major neurological improvement of 8 or more points, or return to the National Institutes of Health Stroke Scale (NIHSS) total score of 0 or 1 at 24 hour(s). | 24 hours
  Early major neurological improvement of 8 or more points, or return to the National Institutes of Health Stroke Scale (NIHSS) total score of 0 or 1 at 24 hour(s).
Health Related Quality of Life (EuroQol five dimensions questionnaire, EQ-5D) | Day 90 (+/- 7)
  Health Related Quality of Life (EuroQol five dimensions questionnaire, EQ-5D)
Barthel Index score | Day 90 (+/- 7)
  Barthel Index score
Need for thrombectomy | 24 hours
  Need for thrombectomy

OTHER OUTCOMES:
Mortality | Day 90 (+/- 7)
  Mortality
Imaging scan up to 36 hours, combined with a neurological deterioration NIHSS≥4 points from baseline (or lowest NIHSS value baseline-24 h), or leading to death (Safe Implementation of Thrombolysis in Stroke-Monitoring study definition). | 36 hours
  Imaging scan up to 36 hours, combined with a neurological deterioration NIHSS≥4 points from baseline (or lowest NIHSS value baseline-24 h), or leading to death (Safe Implementation of Thrombolysis in Stroke-Monitoring study definition).
Symptomatic Intra-Cerebral Haemorrhage (SICH) by (European Cooperative Acute Stroke Study) ECASS-2 and ECASS-3 definitions. | up to day 90
  Symptomatic Intra-Cerebral Haemorrhage (SICH) by (European Cooperative Acute Stroke
Parenchymal Haematoma type 2 (PH2) haemorrhage on post-treatment computerised tomography (CT) scan up to 36 hours after treatment. | 36 hours
  Parenchymal Haematoma type 2 (PH2) haemorrhage on post-treatment computerised
Intracranial haemorrhage | 22-36 hours
  Any intracranial haemorrhage on 22-36 hours computerised tomography (CT) scan
Significant extracranial haemorrhage (requirement for blood transfusion or drop in haemoglobin of ≥20mg/l in the 36h after treatment). | 36 hours
  Significant extracranial haemorrhage (requirement for blood transfusion or drop in haemoglobin of ≥20mg/l in the 36h after treatment).

CONTACTS AND LOCATIONS:
Overall Officials: Keith Muir, MD, FRCP, Principal Investigator — University of Glasgow
Locations (1):
- Queen Elizabeth University Hospital, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Muir KW, Ford GA, Ford I, Wardlaw JM, McConnachie A, Greenlaw N, Mair G, Sprigg N, Price CI, MacLeod MJ, Dima S, Venter M, Zhang L, O'Brien E, Sanyal R, Reid J, Sztriha LK, Haider S, Whiteley WN, Kennedy J, Perry R, Lakshmanan S, Chakrabarti A, Hassan A, Marigold R, Raghunathan S, Sims D, Bhandari M, Wiggam I, Rashed K, Douglass C; ATTEST-2 Investigators. Tenecteplase versus alteplase for acute stroke within 4.5 h of onset (ATTEST-2): a randomised, parallel group, open-label trial. Lancet Neurol. 2024 Nov;23(11):1087-1096. doi: 10.1016/S1474-4422(24)00377-6. PMID 39424558